CLINICAL TRIAL: NCT04917874
Title: Open Label Treatment of Beremagene Geperpavec (B-VEC)
Brief Title: A Long-term Treatment With B-VEC for Dystrophic Epidermolysis Bullosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-VEC-EX-02
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Dystrophic Epidermolysis Bullosa; DEB - Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa; Dominant Dystrophic Epidermolysis Bullosa
Keywords: DEB; Krystal Biotech
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- B-VEC (Experimental): Open label B-VEC topical treatment of DEB wounds.
  Interventions: Biological: Open Label Topical Beremagene Geperpavec (B-VEC)

INTERVENTIONS:
Biological: Open Label Topical Beremagene Geperpavec (B-VEC) — Topical gel of non-integrating, replication-incompetent HSV-1 expressing the human collagen VII protein

SUMMARY:
This is a 112-week (approximately two-year) open-label extension study of Beremagene Geperpavec (B-VEC), for participants aged 2 months and older, who have been diagnosed with Dystrophic Epidermolysis Bullosa (DEB). Participants will be dosed weekly with the topical B-VEC therapy. The primary endpoint will be to assess long term safety and tolerability of the topical gene therapy. The study is for those who participated in Phase 3 study, as well as, new participants who were unable to participate in the Phase 3 study, who meet all enrollment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give consent/assent
* Clinical diagnosis of epidermolysis bullosa
* Confirmation of diagnosis (either DDEB or RDEB) by genetic testing including COL7A1.
* Age: 2 months of age and older at the time of informed consent/assent
* Women of childbearing age must be willing to use reliable birth control method throughout the treatment duration and for 3 months following the last treatment application

Exclusion Criteria:

* Diseases or conditions that could interfere with the assessment of safety of the study treatment and compliance of the participant with study visits/procedures, as determined by the Investigator
* Pregnant or nursing women
* Active infection in the area that will undergo administration, that the Investigator believes will negatively impact the IP application
* Known allergy to any of the constituents of the product
* Concurrent skin transplant or mesh skin grafting; if the participant is currently having transplantation or grafting surgeries they must wait until the transplant has begun to heal and the graft has absorbed prior to initiating B-VEC therapy
* Participation in an interventional gene therapy clinical trial within the past three (3) months (not including B-VEC administration)

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
To record safety outcomes of participants while on B-VEC. | Up to 112 weeks
  Record reportable Adverse (AE) and Serious Adverse Events (SAEs) during the continued use of B-VEC to participants who have participated in and completed Krystal Biotech's Phase 3 Protocol (A Phase 3 Efficacy and Safety Study of Beremagene Geperpavec (B-VEC, previously KB103) for the Treatment of Dystrophic Epidermolysis Bullosa (DEB)), as an extension of use, upon study completion; as well as, for participants diagnosed with DEB who have not participated in the B-VEC Phase 3 trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Chien, MD, Study Director — Senior Vice President of Clinical Development
Locations (6):
- United States (6):
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - Stanford University, Redwood City, California
  - Pediatric Skin Research, Coral Gables, Florida
  - Northwestern University, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ascension Seton- Dell's Children Medical Group, Austin, Texas

REFERENCES:
- [Derived] Marinkovich MP, Paller AS, Guide SV, Gonzalez ME, Lucky AW, Bagci IS, Agostini B, Fitzgerald K, Chen S, Chen H, Conner MM, Krishnan SM. Long-Term Safety and Tolerability of Beremagene Geperpavec-svdt (B-VEC) in an Open-Label Extension Study of Patients with Dystrophic Epidermolysis Bullosa. Am J Clin Dermatol. 2025 Jul;26(4):623-635. doi: 10.1007/s40257-025-00942-y. Epub 2025 Apr 12. PMID 40220208